CLINICAL TRIAL: NCT02223182
Title: A Double-Blind, Placebo-Controlled Randomized Trial to Study the Viaskin Milk Efficacy and Safety for Treating IgE-Mediated Cow's Milk Allergy in Children
Brief Title: Efficacy and Safety of Viaskin Milk in Children With IgE-Mediated Cow's Milk Allergy
Acronym: MILES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MILES
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Food Allergy
Keywords: Milk Allergy,; Viaskin Milk,; Specific Immunotherapy,; Epicutaneous ImmunoTherapy (EPIT); IgE-Mediated Cow's Milk Allergy
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Viaskin Milk 150 mcg (Experimental): One Viaskin epicutaneous delivery system (patch) containing 150µg of cow's milk proteins applied each day for 12 months.
  Interventions: Biological: Viaskin Milk 150 mcg
- Viaskin Milk 300 mcg (Experimental): One Viaskin epicutaneous delivery system (patch) containing 300µg of cow's milk proteins applied each day for 12 months.
  Interventions: Biological: Viaskin Milk 300 mcg
- Viaskin Milk 500 mcg (Experimental): One Viaskin epicutaneous delivery system (patch) containing 500µg of cow's milk proteins applied each day for 12 months.
  Interventions: Biological: Viaskin Milk 500 mcg
- Viaskin Placebo (Placebo Comparator): One Viaskin epicutaneous delivery system (patch) containing placebo applied each day for 12 months.
  Interventions: Biological: Viaskin Placebo

INTERVENTIONS:
Biological: Viaskin Milk 150 mcg — Subjects epicutaneously administered daily (up to 24 hours application per day) with a patch containing 150 mcg cow's milk proteins.
  Arms: Viaskin Milk 150 mcg
Biological: Viaskin Milk 300 mcg — Subjects epicutaneously administered daily (up to 24 hours application per day) with a patch containing 300 mcg cow's milk proteins.
  Arms: Viaskin Milk 300 mcg
Biological: Viaskin Milk 500 mcg — Subjects epicutaneously administered daily (up to 24 hours application per day) with a patch containing 500 mcg cow's milk proteins.
  Arms: Viaskin Milk 500 mcg
Biological: Viaskin Placebo — Subjects epicutaneously administered daily (up to 24 hours application per day) with a patch containing a matching placebo formulation.
  Arms: Viaskin Placebo

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of Viaskin Milk after 12 months of epicutaneous immunotherapy (EPIT) treatment, for desensitizing IgE-mediated cow's milk allergic children and to assess the long-term safety and therapeutic benefit with Viaskin Milk.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, placebo-controlled, randomized trial to study the safety and efficacy of Viaskin Milk applied epicutaneously every day to subjects from 2 to 17 years of age with IgE-mediated cow's milk allergy (CMA). Subjects will receive blinded treatment for 1 year at one of the 3 doses of Viaskin Milk: 150µg, 300µg, 500µg or placebo. After the first year, all subjects were to switch to the highest dose of Viaskin Milk, 500µg, and continue treatment in an open-label manner for up to a maximum of 3 additional years. Following results of the 12-month blinded period, all eligible subjects who wish to continue participation in the study will switch from Viaskin Milk 500µg to Viaskin Milk 300µg for 24 months of treatment.

Eligible subjects with confirmed IgE-mediated CMA will perform a first Double-Blind Placebo-Controlled Food Challenge (DBPCFC) at screening with escalating doses of cow's milk proteins. Subjects showing a positive DBPCFC at screening, defined as the appearance of objective signs or symptoms to an eliciting dose of cow's milk proteins ≤300 mg (approximately ≤9.4mL of cow's milk) will be randomized in the study to receive a 12 month treatment (blinded treatment period), at which time a second DBPCFC will be performed to evaluate the primary efficacy endpoint of the study.

Approximately 194 subjects will be randomized in this study. The total duration of participation in the study will differ for each individual subject and could be up to approximately 6 years.

ELIGIBILITY:
Eligibility criteria for study enrollment:

Inclusion Criteria:

* Signed Informed Consent Form (ICF) by parent(s)/guardian(s) of subjects and informed assent form (IAF) for subjects ≥7 years, or as per local or country specific guidelines or regulations.
* Male or female subjects 2 to 17 years old at Visit 1.
* Documented medical history or physician-confirmed diagnosis of IgE-mediated CMA with systemic symptoms related to ingestion of milk or dairy products.
* Subjects currently following a strict cow's milk-free diet, with no consumption of dairy or baked milk products.
* Cow's milk-specific IgE level at screening ≥10 kU/L
* Positive Skin Prick Test (SPT) to cow's milk with a largest wheal diameter ≥6 mm.
* Positive DBPCFC at screening with an eliciting dose ≤300 mg cow's milk proteins (approximately ≤9.4 mL of cow's milk).
* Negative urine pregnancy test for female subjects of childbearing potential. Female subjects of childbearing potential must agree and commit to use effective medical methods of contraception for the entire duration of their participation in the study. Sexual abstinence will be accepted as an effective method of contraception for girls below 15 years of age.
* Ability to perform spirometry procedures in accordance with the American Thoracic Society guidelines (2005) for subjects ≥6 years old. Ability to perform peak expiratory flow (PEF) measurements for subjects ≥5 years old. Subjects <8 years of age who have documented inability to adequately perform spirometry can perform only the PEF evaluation. Subjects <5 years of age may be enrolled if they had no clinical features of moderate or severe persistent asthma severity (as defined by the 2007 National Heart, Lung, and Blood Institute [NHLBI] Guidelines) within 1 year before Visit 1.
* Subjects and/or parents/guardians willing to comply with all study requirements during participation in the study.

Exclusion Criteria:

* History of severe anaphylaxis to cow's milk resulting in hypotension, hypoxia or neurological compromise (collapse, loss of consciousness or incontinence) or requiring mechanical ventilation.
* Pregnancy or lactation.
* Spirometry forced expiratory volume in 1 second (FEV1) <80% of the predicted value at Visit 1 for subjects ≥6 years and able to perform the spirometry, or PEF <80% of predicted value at Visit 1 for subjects performing only the PEF measurements.
* Any clinical features of moderate or severe persistent asthma severity (as defined by the 2007 NHLBI guidelines) and high daily doses of inhaled corticosteroids.
* Known allergy to the Viaskin patch materials or excipients, or to any of the components of the food challenge formulas other than the cow's milk proteins.
* Allergy or known history of reaction to Tegaderm® medical dressing with no possibility to use an alternative adhesive dressing authorized by the sponsor in replacement.
* Subjects having objective symptoms to the placebo formula leading to stopping the challenge during the screening DBPCFC.
* Severe reaction during the screening DBPCFC defined as need for intubation, and/or hypotension persisting after epinephrine administration, and/or the need for >2 doses of epinephrine.
* Symptomatic allergy to pollens with symptoms during the pollen season that might interfere with the symptoms observed during the DBPCFC, if the DBPCFC is performed during the pollen season. Screening of such subjects should be made out of the pollen season.
* Inability to discontinue short-acting antihistamines for 3 days or long-acting antihistamines for 5 to 7 days (depending on the half-life) before the DBPCFC.
* Use of systemic long-acting corticosteroids within 12 weeks before Visit 1 and/or use of systemic short-acting corticosteroids within 4 weeks before Visit 1 or use of systemic long-acting or short-acting corticosteroids during screening (unless used to treat symptoms triggered by the DBPCFC or triggered by accidental allergen consumption; in the latter case DBPCFC must then be scheduled after a minimum of 7 wash-out days).
* Subjects with asthma conditions meeting 1 or several criteria below:

  * Uncontrolled persistent asthma (as defined by the 2007 NHLBI guidelines) or subject being treated with a combination therapy of medium or high daily dose of inhaled corticosteroid with a long acting inhaled β2-agonist. Intermittent asthmatic subjects who require intermittent use of inhaled corticosteroids for rescue are permitted.
  * At least 2 systemic corticosteroid courses for asthma within 1 year before Visit 1 or 1 oral corticosteroid course for asthma within 3 months before Visit 1, or during screening (unless used to treat symptoms triggered by the DBPCFC).
  * Prior intubation/mechanical ventilation due to asthma within 2 years before Visit 1, or during screening.
* Upper respiratory infection or gastroenteritis within 7 days of DBPCFC (DBPCFC must then be rescheduled at least 7 days after resolution of these conditions).
* Any history of milk immunotherapy (eg, oral immunotherapy, sublingual immunotherapy or specific oral tolerance induction).
* Prior history of any other food allergen immunotherapy (eg, oral immunotherapy, sublingual immunotherapy or specific oral tolerance induction) within 5 years before Visit 1.
* Subjects currently under aeroallergen immunotherapy and unwilling or unable to discontinue at the time of Visit 1. Aeroallergen Immunotherapy must be discontinued at the time of Visit 1.
* Use of any anti-IgE drug (eg, omalizumab), any immunomodulatory therapy, or any biological agent therapy (eg, anti-tumor necrosis factor drugs) within 1 year before Visit 1, or during screening.
* Generalized dermatologic diseases (eg, severe atopic dermatitis, uncontrolled generalized eczema, icthyosis vulgaris) with no intact zones to apply the Viaskin patch, or urticarial and mast cells disorders such as chronic idiopathic urticaria.
* Subject and/or subject's parents/guardians with obvious excessive anxiety and unlikely to cope with the conditions of a food challenge.
* Past or current disease, including but not limited to active eosinophilic gastrointestinal disorders, autoimmune disorders, immunodeficiency, malignancy, uncontrolled disease (hypertension, diabetes, psychiatric disorder, cardiac disease), or other disorders (eg, liver, gastrointestinal, kidney, cardiovascular, pulmonary disease or blood disorder) which in the opinion of the Investigator or the sponsor may affect the subject's participation in the study or place the subject at increased risk.
* Subjects and/or parents/guardians unable to use the epinephrine auto-injector properly in spite of being adequately trained.
* Contraindicated condition for the use of epinephrine.
* Use of any investigational drug or device, or participation in another interventional clinical study within 3 months before Visit 1.
* Subjects receiving beta-blockers or Angiotensin converting-enzyme (ACE) inhibitors.
* Subjects unable to follow the protocol requirements.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (12):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rady Children's Hospital, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - ASTHMA, Inc., Seattle, Washington
- Canada (5):
  - Cheema Research Inc., Mississauga, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec
  - Clinique Spécialisée en allergie de la Capitale, Québec

REFERENCES:
- [Derived] Petroni D, Begin P, Bird JA, Brown-Whitehorn T, Chong HJ, Fleischer DM, Gagnon R, Jones SM, Leonard S, Makhija MM, Oriel RC, Shreffler WG, Sindher SB, Sussman GL, Yang WH, Bee KJ, Bois T, Campbell DE, Green TD, Rutault K, Sampson HA, Wood RA. Varying Doses of Epicutaneous Immunotherapy With Viaskin Milk vs Placebo in Children With Cow's Milk Allergy: A Randomized Clinical Trial. JAMA Pediatr. 2024 Apr 1;178(4):345-353. doi: 10.1001/jamapediatrics.2023.6630. PMID 38407859

RESULTS

PARTICIPANT FLOW:
Period: Double-Blind Period
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Started | 49 | 49 | 47 | 53
Completed | 47 | 45 | 45 | 52
Not Completed | 2 | 4 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Non Compliance | 0 | 0 | 0 | 1
Not completed — Sponsor or Regulatory Authorities Decision | 1 | 0 | 0 | 0
Period: Open-Label 500 Period
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Started | 46 | 45 | 44 | 52
Completed | 40 | 43 | 32 | 42
Not Completed | 6 | 2 | 12 | 10
Not completed — Adverse Event | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 9 | 8
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Sponsor or Regulatory Authorities Decision | 0 | 0 | 1 | 0
Period: Open-Label 300 Period
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Started | 34 | 38 | 29 | 39
Completed | 23 | 23 | 14 | 24
Not Completed | 11 | 15 | 15 | 15
Not completed — Withdrawal by Subject | 10 | 13 | 13 | 15
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Non Compliance | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall Intent-to-Treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo | Total
Number analyzed (Participants) | 49 | 49 | 47 | 53 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (4.56) | 7.7 (4.34) | 8.7 (3.37) | 8.1 (4.31) | 8.0 (4.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 12 | 20 | 18 | 74
  Male | 25 | 37 | 27 | 35 | 124
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 33 | 28 | 31 | 41 | 133
  Black | 1 | 2 | 4 | 1 | 8
  Hispanic | 2 | 1 | 1 | 1 | 5
  Asian | 8 | 10 | 9 | 5 | 32
  Other | 5 | 8 | 2 | 5 | 20
Skin Prick Test Mean wheal diameter [Median (Inter-Quartile Range); unit: millimeters] — Skin Prick Test Mean wheal diameter to Cow's milk
  millimeters | 10.5 [9.0 to 12.0] | 11.0 [9.0 to 13.5] | 10.5 [9.5 to 13.8] | 11.0 [9.0 to 14.5] | 10.5 [9.0 to 13.5]
Cumulative Reactive Dose (CRD) of Cow's milk [Median (Inter-Quartile Range); unit: mg of cow's milk proteins] — Cumulative Reactive Dose of Cow's Milk proteins during the screening Double-Blind Placebo-Controlled Food Challenge
  mg of cow's milk proteins | 144 [44 to 444] | 144 [44 to 444] | 144 [44 to 444] | 144 [44 to 444] | 144 [44 to 444]
Cow's milk sIgE [Median (Inter-Quartile Range); unit: kU/L] | 58.2 [31.5 to 115] | 67.6 [31.0 to 187.0] | 64.6 [32.1 to 291.0] | 61.1 [24.8 to 163.0] | 61.9 [31.5 to 163]
Cow's milk sIgG4 [Median (Inter-Quartile Range); unit: mgA/L] | 14.0 [11.5 to 17.1] | 14.5 [12.3 to 16.4] | 14.0 [12.7 to 16.3] | 13.5 [11.9 to 16.9] | 14.0 [12.0 to 16.9]

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Subjects Who Are Treatment Responders After 12 Months of EPIT Treatment.
Description: A treatment responder is defined as a subject who meets at least one of the following criteria:
  * A ≥10-fold increase in the Cumulative Reactive Dose (CRD) of cow's milk proteins at the Month 12 double-blind placebo-controlled food challenge (DBPCFC) as compared to baseline value and reaching at least 144 mg of cow's milk proteins;
  * A CRD of cow's milk proteins ≥1444 mg at the Month 12 DBPCFC.
Time Frame: From baseline to Month 12 (double-blind period)
Population: Overall Intent-to-Treat Population
Measure: Number; unit: percent of participants
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 49 | 49 | 47 | 53
percent of participants | 36.7 | 49.0 | 36.2 | 30.2

2. Secondary Outcome: Mean Cumulative Reactive Dose (CRD) of Cow's Milk Proteins.
Description: Change in CRD from Month 0 (baseline) to Month 12 Double-Blind Placebo-Controlled Food Challenge expressed in mg of cow's milk proteins.
Time Frame: From baseline to Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Mean (Standard Deviation); unit: milligrams (mg) of cow's milk proteins
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 48 | 45 | 45 | 52
milligrams (mg) of cow's milk proteins | 745.1 (1197.08) | 1201.0 (1675.90) | 723.5 (1218.26) | 555.5 (1143.21)

3. Secondary Outcome: Median Cumulative Reactive Dose (CRD) of Cow's Milk Proteins.
Description: Change in Median CRD from Month 0 (baseline) to Month 12 Double-Blind Placebo-Controlled Food Challenge expressed in mg of cow's milk proteins.
Time Frame: From baseline to Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: milligrams (mg) of cow's milk proteins
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 48 | 45 | 45 | 52
milligrams (mg) of cow's milk proteins | 300 [3 to 1145] | 400 [100 to 1325] | 93 [0 to 1300] | 100 [0 to 900]

4. Secondary Outcome: Change in Levels of sIgE to Cow's Milk.
Description: Median change from baseline value in levels of IgE specific to cow's milk proteins
Time Frame: From baseline to Week 3, Month 3, Month 6, Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: kU/L
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 48 | 49 | 47 | 53
kU/L
  Week 3 | -2.43 [-15.75 to 8.20] | 2.80 [-3.90 to 17.10] | -2.30 [-11.40 to 11.70] | -5.40 [-28.00 to 1.10]
  Month 3: number analyzed (Participants) | 48 | 47 | 44 | 53
  Month 3 | -0.70 [-18.20 to 11.90] | 3.20 [-10.00 to 27.00] | -6.99 [-20.75 to 7.10] | -7.20 [-28.50 to 0.90]
  Month 6: number analyzed (Participants) | 47 | 47 | 44 | 52
  Month 6 | -5.80 [-37.80 to 3.80] | -5.00 [-19.40 to 6.00] | -14.40 [-54.95 to 2.70] | -5.45 [-31.30 to 4.25]
  Month 12: number analyzed (Participants) | 47 | 45 | 45 | 53
  Month 12 | -5.90 [-40.50 to 7.30] | -2.70 [-16.10 to 13.30] | -20.60 [-69.00 to -6.00] | -7.70 [-27.70 to 1.80]

5. Secondary Outcome: Change in Levels of sIgG4 to Cow's Milk.
Description: Median change from baseline value in levels of IgG4 specific to cow's milk proteins
Time Frame: From baseline to Week 3, Month 3, Month 6, Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: mgA/L
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 49 | 49 | 47 | 53
mgA/L
  Week 3: number analyzed (Participants) | 49 | 49 | 47 | 52
  Week 3 | 0.24 [-1.74 to 2.00] | 0.90 [-1.30 to 2.80] | 0.80 [-0.70 to 2.70] | -0.35 [-2.10 to 1.89]
  Month 3: number analyzed (Participants) | 48 | 46 | 43 | 53
  Month 3 | 0.90 [-0.75 to 2.45] | 2.45 [0.10 to 4.50] | 2.60 [-1.60 to 5.90] | -0.80 [-2.60 to 1.00]
  Month 6: number analyzed (Participants) | 47 | 47 | 44 | 53
  Month 6 | 0.10 [-2.00 to 3.29] | 1.30 [-1.20 to 5.00] | 1.40 [-1.70 to 5.75] | -1.60 [-3.10 to 0.40]
  Month 12: number analyzed (Participants) | 49 | 45 | 45 | 53
  Month 12 | 1.20 [-1.40 to 4.10] | 3.50 [-0.50 to 10.00] | 1.96 [-0.20 to 11.80] | -1.60 [-2.74 to -0.30]

6. Secondary Outcome: Change in Levels of sIgE to Caseins, α-lactalbumin and β-lactoglobulin
Description: Median change from baseline in levels of IgE specific to caseins, α-lactalbumin and β-lactoglobulin proteins
Time Frame: From baseline to Week 3, Month 3, Month 6, Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: kU/L
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 48 | 49 | 47 | 53
kU/L
  Caseins - Week 3: number analyzed (Participants) | 48 | 49 | 47 | 52
  Caseins - Week 3 | -2.09 [-14.80 to 4.44] | 0.15 [-5.00 to 19.00] | 0.50 [-8.50 to 10.70] | -1.80 [-7.75 to 6.10]
  Caseins - Month 3: number analyzed (Participants) | 48 | 47 | 44 | 53
  Caseins - Month 3 | 1.15 [-20.35 to 11.49] | -0.20 [-9.50 to 27.20] | 1.15 [-8.95 to 11.45] | -2.46 [-14.70 to 10.00]
  Caseins - Month 6: number analyzed (Participants) | 47 | 47 | 44 | 52
  Caseins - Month 6 | -5.60 [-38.40 to 4.98] | -5.80 [-31.00 to 6.10] | -8.45 [-46.50 to 3.10] | -2.55 [-17.75 to 5.50]
  Caseins - Month 12: number analyzed (Participants) | 47 | 45 | 45 | 53
  Caseins - Month 12 | -5.80 [-32.40 to 1.58] | -2.00 [-29.00 to 2.90] | -12.60 [-92.00 to -1.20] | -4.45 [-16.30 to 7.90]
  α-lactalbumin - Week 3 | 0.07 [-2.18 to 2.50] | -0.06 [-1.89 to 4.10] | -0.10 [-3.20 to 2.60] | -0.48 [-3.00 to 0.46]
  α-lactalbumin - Month 3: number analyzed (Participants) | 48 | 47 | 44 | 53
  α-lactalbumin - Month 3 | -0.16 [-4.35 to 1.31] | 0.18 [-2.90 to 5.20] | -1.78 [-5.70 to 0.40] | -1.00 [-2.84 to 0.90]
  α-lactalbumin - Month 6: number analyzed (Participants) | 47 | 47 | 44 | 52
  α-lactalbumin - Month 6 | -1.21 [-7.88 to 0.51] | -0.53 [-3.93 to 3.80] | -3.72 [-13.10 to -0.03] | -0.71 [-4.41 to 0.60]
  α-lactalbumin - Month 12: number analyzed (Participants) | 47 | 45 | 45 | 53
  α-lactalbumin - Month 12 | -4.60 [-11.30 to 0.09] | -1.76 [-9.30 to 0.05] | -7.20 [-18.90 to -1.10] | -1.20 [-6.50 to 0.00]
  β-lactoglobulin - Week 3 | -0.04 [-2.45 to 0.71] | 0.45 [-0.54 to 3.79] | 0.00 [-2.07 to 3.23] | -0.41 [-3.30 to 0.33]
  β-lactoglobulin - Month 3: number analyzed (Participants) | 48 | 47 | 44 | 53
  β-lactoglobulin - Month 3 | -0.02 [-2.25 to 1.06] | 1.40 [-1.60 to 6.00] | -1.17 [-3.46 to 0.55] | -0.60 [-3.33 to 1.54]
  β-lactoglobulin - Month 6: number analyzed (Participants) | 47 | 47 | 44 | 52
  β-lactoglobulin - Month 6 | -0.29 [-7.40 to 0.06] | -0.12 [-4.02 to 6.10] | -3.55 [-11.83 to -0.02] | -1.11 [-5.52 to 0.24]
  β-lactoglobulin - Month 12: number analyzed (Participants) | 47 | 45 | 45 | 53
  β-lactoglobulin - Month 12 | -1.36 [-11.00 to -0.24] | -0.92 [-7.33 to 0.58] | -4.02 [-14.50 to -1.63] | -2.29 [-7.00 to -0.01]

7. Secondary Outcome: Change in Levels of sIgG4 to Caseins, α-lactalbumin and β-lactoglobulin
Description: Median change from baseline in levels of IgG4 specific to caseins, α-lactalbumin and β-lactoglobulin proteins
Time Frame: From baseline to Week 3, Month 3, Month 6, Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: mgA/L
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 49 | 49 | 47 | 53
mgA/L
  Caseins - Week 3: number analyzed (Participants) | 49 | 49 | 47 | 52
  Caseins - Week 3 | 0.11 [-0.06 to 0.25] | 0.15 [-0.07 to 1.05] | 0.15 [-0.14 to 1.19] | 0.03 [-0.22 to 0.17]
  Caseins - Month 3: number analyzed (Participants) | 48 | 47 | 43 | 53
  Caseins - Month 3 | 0.39 [0.00 to 0.99] | 1.08 [0.31 to 2.66] | 0.78 [0.11 to 2.00] | -0.06 [-0.35 to 0.14]
  Caseins - Month 6: number analyzed (Participants) | 47 | 46 | 44 | 53
  Caseins - Month 6 | 0.32 [0.14 to 1.64] | 1.04 [0.20 to 2.69] | 0.69 [0.19 to 1.75] | -0.01 [-0.37 to 0.14]
  Caseins - Month 12: number analyzed (Participants) | 49 | 45 | 45 | 53
  Caseins - Month 12 | 0.47 [-0.18 to 1.47] | 1.05 [0.04 to 2.73] | 0.61 [0.10 to 4.43] | -0.11 [-0.51 to 0.17]
  α-lactalbumin - Week 3: number analyzed (Participants) | 49 | 49 | 47 | 52
  α-lactalbumin - Week 3 | 0.00 [-0.07 to 0.17] | 0.06 [-0.01 to 0.43] | 0.00 [-0.05 to 0.65] | 0.00 [-0.08 to 0.09]
  α-lactalbumin - Month 3: number analyzed (Participants) | 48 | 47 | 43 | 53
  α-lactalbumin - Month 3 | 0.63 [0.22 to 1.19] | 0.81 [0.23 to 2.04] | 0.65 [0.00 to 2.32] | 0.00 [-0.05 to 0.13]
  α-lactalbumin - Month 6: number analyzed (Participants) | 47 | 46 | 44 | 53
  α-lactalbumin - Month 6 | 1.09 [0.25 to 2.20] | 1.64 [0.62 to 2.80] | 1.19 [0.08 to 3.48] | 0.00 [-0.04 to 0.13]
  α-lactalbumin - Month 12: number analyzed (Participants) | 49 | 45 | 45 | 53
  α-lactalbumin - Month 12 | 1.28 [0.52 to 3.48] | 2.72 [0.74 to 7.38] | 1.94 [0.46 to 6.46] | 0.00 [-0.18 to 0.08]
  β-lactoglobulin - Week 3: number analyzed (Participants) | 49 | 49 | 47 | 52
  β-lactoglobulin - Week 3 | 0.03 [-0.01 to 0.24] | 0.08 [-0.03 to 0.29] | 0.11 [-0.02 to 0.61] | 0.00 [-0.10 to 0.07]
  β-lactoglobulin - Month 3: number analyzed (Participants) | 48 | 47 | 43 | 53
  β-lactoglobulin - Month 3 | 0.22 [0.01 to 1.00] | 0.67 [0.35 to 1.73] | 0.65 [0.12 to 2.11] | -0.01 [-0.21 to 0.13]
  β-lactoglobulin - Month 6: number analyzed (Participants) | 47 | 46 | 44 | 53
  β-lactoglobulin - Month 6 | 0.36 [0.04 to 1.20] | 0.94 [0.33 to 2.37] | 0.88 [0.06 to 2.30] | -0.03 [-0.20 to 0.11]
  β-lactoglobulin - Month 12: number analyzed (Participants) | 49 | 45 | 45 | 53
  β-lactoglobulin - Month 12 | 0.47 [0.09 to 2.17] | 2.06 [0.63 to 4.78] | 1.55 [0.23 to 3.33] | -0.06 [-0.27 to 0.03]

8. Secondary Outcome: Change in Skin Prick Test (SPT) Wheal.
Description: Median change from baseline in SPT Wheal diameter
Time Frame: From baseline to Month 3, Month 6, Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: millimeters (mm)
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 48 | 47 | 46 | 52
millimeters (mm)
  Month 3: number analyzed (Participants) | 48 | 45 | 46 | 52
  Month 3 | -1 [-3 to 2] | -1 [-4 to 2] | -1 [-3 to 2] | 0 [-3 to 4]
  Month 6: number analyzed (Participants) | 48 | 47 | 42 | 51
  Month 6 | 0 [-3 to 3] | -2 [-4 to 1] | -1 [-4 to 1] | 0 [-4 to 3]
  Month 12: number analyzed (Participants) | 48 | 45 | 45 | 52
  Month 12 | 0 [-4 to 3] | -1 [-4 to 1] | -1 [-3 to 2] | 0 [-3 to 2]

9. Secondary Outcome: Change in the Severity of Symptoms Elicited During the Milk Double-Blind Placebo-Controlled Food Challenge (DBPCFC).
Description: Summary of total objective severity score for DBPCFC. The total objective severity score is calculated as the sum of the severity grades (0-Absent, 1-Mild, 2-Moderate or 3-Severe) of the following objective symptoms: pruritus, urticaria/angioedema, rash, sneezing/itching, nasal congestion, rhinorrhea, laryngeal, wheezing, diarrhea, vomiting, cardiovascular and conjunctivitis for DBPCFC with cow's milk formula.
  The total objective score ranges from a minimum of 0 to a maximum of 36 (if the maximum grade 3 was reported for each of the 12 symptoms), with a higher score meaning a worse outcome. A negative score in the changes to Month 0 means improvement.
Time Frame: From baseline to Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 49 | 49 | 47 | 53
score on a scale
  Month 0 | 6 [4 to 9] | 6 [4 to 8] | 6 [4 to 10] | 6 [4 to 9]
  Month 12: number analyzed (Participants) | 48 | 45 | 45 | 52
  Month 12 | 5 [4 to 9] | 6 [3 to 9] | 6 [4 to 9] | 6 [3 to 10]
  Change from Month 0 to Month 12: number analyzed (Participants) | 48 | 45 | 45 | 52
  Change from Month 0 to Month 12 | -1 [-3 to 3] | 0 [-2 to 2] | 0 [-2 to 2] | 0 [-3 to 3]

10. Secondary Outcome: Change in Quality of Life (QoL) Assessments.
Description: Summary of Global Score for Food Allergy Quality of Life Questionnaire Parent Child Form (FAQLQ-PF). The scores range from 1 (no problem/impairment) to 7 (maximal problem/impairment). A negative score in the changes to Month 0 means improvement.
Time Frame: From baseline to Month 12 (double-blind period)
Population: All subjects from the Intent-to-Treat population for whom this outcome measure was collected and analyzed
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 39 | 39 | 41 | 44
score on a scale
  Month 0 | 4.6 [3.3 to 5.4] | 4.4 [3.4 to 5.2] | 4.6 [3.6 to 5.2] | 4.9 [3.3 to 5.5]
  Month 12: number analyzed (Participants) | 39 | 38 | 39 | 44
  Month 12 | 4.3 [3.4 to 5.2] | 4.5 [3.5 to 5.4] | 4.3 [3.7 to 5.1] | 4.1 [3.4 to 5.2]
  Change from Month 0 to Month 12: number analyzed (Participants) | 39 | 38 | 39 | 44
  Change from Month 0 to Month 12 | -0.1 [-0.6 to 0.5] | 0.1 [-0.2 to 0.5] | 0 [-0.8 to 0.5] | -0.4 [-0.8 to 0.5]

11. Secondary Outcome: Percentage (%) of Subjects Who Are Treatment Responders Over the Course of the Viaskin Milk 300µg Open-label Treatment Period Using Observed Data
Description: A treatment responder is defined as a subject who meets at least one of the following criteria:
  A ≥10-fold increase in the Cumulative Reactive Dose (CRD) of cow's milk proteins at the Month 12 double-blind placebo-controlled food challenge (DBPCFC) as compared to baseline value and reaching at least 144 mg of cow's milk proteins; A CRD of cow's milk proteins ≥1444 mg at the Month 12 DBPCFC.
  DBPCFC at Month 12 and Month 24 after switch to Viaskin Milk 300µg was optional and therefore outcome measure was assessed on observed data only.
Time Frame: From baseline to Month 12 and Month 24 after switch to Viaskin Milk 300µg (Open-Label 300µg period)
Population: All subjects from the Open-Label Set 300 (OLS-300) for whom this outcome measure was collected and analyzed. OLS-300 includes all subjects who entered the open-label treatment period after switch to Viaskin Milk 300µg and applied at least one Viaskin Milk 300µg patch during this open-label period.
Measure: Number; unit: Percentage of participants
Groups:
- Viaskin Milk 150 mcg: One Viaskin epicutaneous delivery system (patch) containing 150µg of cow's milk proteins applied each day for 12 months (double-blind period), followed by a patch containing 500µg of cow's milk proteins (Open-label 500µg period), followed by a patch containing 300µg for up to 24 months (Open-label 300µg period).
  One patch applied each day (up to 24 hours) during the double-blind and open-label periods.
- Viaskin Milk 300 mcg: One Viaskin epicutaneous delivery system (patch) containing 300µg of cow's milk proteins applied each day for 12 months (double-blind period), followed by a patch containing 500µg of cow's milk proteins (Open-label 500µg period), followed by a patch containing 300µg for up to 24 months (Open-label 300µg period).
  One patch applied each day (up to 24 hours) during the double-blind and open-label periods.
- Viaskin Milk 500 mcg: One Viaskin epicutaneous delivery system (patch) containing 500µg of cow's milk proteins applied each day for 12 months (double-blind period), followed by a patch containing 500µg of cow's milk proteins (Open-label 500µg period), followed by a patch containing 300µg for up to 24 months (Open-label 300µg period).
  One patch applied each day (up to 24 hours) during the double-blind and open-label periods.
- Viaskin Placebo: One Viaskin epicutaneous delivery system (patch) containing placebo applied each day for 12 months (double-blind period), followed by a patch containing 500µg of cow's milk proteins (Open-label 500µg period), followed by a patch containing 300µg for up to 24 months (Open-label 300µg period).
  One patch applied each day (up to 24 hours) during the double-blind and open-label periods.
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 15 | 13 | 8 | 14
Percentage of participants
  Month 12 after switch to Viaskin Milk 300µg: number analyzed (Participants) | 14 | 11 | 8 | 11
  Month 12 after switch to Viaskin Milk 300µg | 85.7 | 72.7 | 62.5 | 81.8
  Month 24 after switch to Viaskin Milk 300µg | 80.0 | 84.6 | 50.0 | 64.3

12. Secondary Outcome: Cumulative Reactive Dose (CRD) of Cow's Milk Protein Over the Course of the Open-label Treatment Period
Description: Median CRD during Double-Blind Placebo-Controlled Food Challenge expressed in mg of cow's milk proteins.
Time Frame: Baseline, Month 12 and Month 24 after switch to Viaskin Milk 300µg (Open-Label 300µg period)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: milligrams (mg) of cow's milk proteins
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 34 | 38 | 29 | 39
milligrams (mg) of cow's milk proteins
  Month 0 | 144 [44 to 444] | 144 [44 to 444] | 144 [44 to 444] | 144 [44 to 444]
  Month 12 after switch to Viaskin Milk 300µg: number analyzed (Participants) | 14 | 11 | 8 | 11
  Month 12 after switch to Viaskin Milk 300µg | 1444 [944 to 6444] | 1444 [444 to 2194] | 1319 [444 to 3481] | 1444 [444 to 6444]
  Month 24 after switch to Viaskin Milk 300µg: number analyzed (Participants) | 15 | 13 | 8 | 14
  Month 24 after switch to Viaskin Milk 300µg | 1444 [474 to 3444] | 1444 [444 to 3444] | 1219 [144 to 2819] | 1444 [444 to 6444]

13. Secondary Outcome: Treatment-Emergent Adverse Events
Description: Overview of Treatment Emergent Adverse Events (TEAEs) and serious Treatment-Emergent Adverse Events
Time Frame: Whole study including double-blind and open-label periods (up to 6 years).
Population: Safety set. It includes all subjects who applied at least one Viaskin patch.
Measure: Number; unit: participants
Arm/Group | Viaskin Milk 150 mcg | Viaskin Milk 300 mcg | Viaskin Milk 500 mcg | Viaskin Placebo
Number analyzed (Participants) | 49 | 49 | 47 | 53
participants
  Any TEAE | 49 | 48 | 47 | 53
  Any serious TEAE | 9 | 6 | 6 | 7
  Any TEAE related to the Investigational Product | 46 | 43 | 39 | 48
  Any serious TEAE related to the Investigational Product | 0 | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected over the entire course of the study including the double-blind period and the open-label periods, up to 6 years overall.
Description: Treatment-Emergent Adverse events during the whole study period.
Groups:
- Double-Blind Viaskin Milk 150 mcg: One Viaskin epicutaneous delivery system (patch) containing 150µg of cow's milk proteins applied each day for 12 months (double-blind period).
- Double-Blind Viaskin Milk 300 mcg: One Viaskin epicutaneous delivery system (patch) containing 300µg of cow's milk proteins applied each day for 12 months (double-blind period).
- Double-Blind Viaskin Milk 500 mcg: One Viaskin epicutaneous delivery system (patch) containing 500µg of cow's milk proteins applied each day for 12 months (double-blind period).
- Double-Blind Viaskin Placebo: One Viaskin epicutaneous delivery system (patch) containing placebo applied each day for 12 months (double-blind period).
- Open-Label Viaskin Milk 500 mcg: One Viaskin epicutaneous delivery system (patch) containing 500µg of cow's milk proteins applied each day for up to 3 years.
  Open-Label Set 500 (OLS-500) that includes all subjects who entered the OL-500 period and applied at least one Viaskin Milk 500µg patch during this Open-Label period (N=185).
- Open-Label Viaskin Milk 300 mcg: One Viaskin epicutaneous delivery system (patch) containing 300µg of cow's milk proteins applied each day for 24 months
  Open-Label Set 300 (OLS-300) that includes all subjects who entered the OL-300 period after switch to Viaskin Milk 300µg and applied at least one Viaskin Milk 300µg patch during this Open-label period (N=140).
Arm/Group | Double-Blind Viaskin Milk 150 mcg | Double-Blind Viaskin Milk 300 mcg | Double-Blind Viaskin Milk 500 mcg | Double-Blind Viaskin Placebo | Open-Label Viaskin Milk 500 mcg | Open-Label Viaskin Milk 300 mcg
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/47 | 0/53 | 0/185 | 0/140
Serious Adverse Events (participants affected / at risk) | 3/49 | 2/49 | 1/47 | 2/53 | 16/185 | 7/140
Other Adverse Events (participants affected / at risk) | 49/49 | 48/49 | 47/47 | 53/53 | 181/185 | 131/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Viaskin Milk 150 mcg (N=49) | Double-Blind Viaskin Milk 300 mcg (N=49) | Double-Blind Viaskin Milk 500 mcg (N=47) | Double-Blind Viaskin Placebo (N=53) | Open-Label Viaskin Milk 500 mcg (N=185) | Open-Label Viaskin Milk 300 mcg (N=140)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Croup Infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road Traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Viaskin Milk 150 mcg (N=49) | Double-Blind Viaskin Milk 300 mcg (N=49) | Double-Blind Viaskin Milk 500 mcg (N=47) | Double-Blind Viaskin Placebo (N=53) | Open-Label Viaskin Milk 500 mcg (N=185) | Open-Label Viaskin Milk 300 mcg (N=140)
Upper respiratory tract infection (Infections and infestations) | 27 (57) | 23 (45) | 16 (32) | 19 (33) | 60 (125) | 38 (73)
Viral upper respiratory tract infection (Infections and infestations) | 11 (24) | 9 (20) | 11 (21) | 10 (21) | 34 (56) | 22 (45)
Influenza (Infections and infestations) | 4 (6) | 3 (4) | 5 (6) | 6 (6) | 29 (29) | 23 (30)
Gastroenteritis viral (Infections and infestations) | 7 (7) | 1 (1) | 3 (4) | 4 (4) | 21 (22) | 10 (12)
Viral infection (Infections and infestations) | 3 (5) | 4 (5) | 4 (5) | 0 (0) | 15 (16) | 20 (35)
Pharyngitis streptococcal (Infections and infestations) | 4 (4) | 3 (3) | 6 (7) | 7 (7) | 15 (22) | 6 (14)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (4) | 1 (1) | 4 (9) | 15 (21) | 9 (11)
Otitis media (Infections and infestations) | 5 (5) | 2 (4) | 4 (4) | 3 (4) | 10 (13) | 1 (4)
Ear infection (Infections and infestations) | 6 (6) | 3 (8) | 1 (1) | 4 (5) | 8 (12) | 5 (10)
Pneumonia (Infections and infestations) | 3 (3) | 1 (2) | 3 (4) | 1 (1) | 10 (13) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 2 (3) | 3 (3) | 10 (10) | 3 (5)
Impetigo (Infections and infestations) | 1 (3) | 1 (2) | 3 (4) | 2 (2) | 4 (4) | 2 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 3 (3) | 5 (5)
Croup infectious (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 29 (129) | 25 (182) | 24 (64) | 16 (45) | 92 (386) | 39 (240)
Application site pruritus (General disorders) | 26 (106) | 26 (128) | 18 (71) | 10 (26) | 86 (395) | 30 (158)
Application site swelling (General disorders) | 14 (78) | 13 (51) | 14 (40) | 3 (7) | 47 (222) | 14 (103)
Pyrexia (General disorders) | 11 (22) | 7 (12) | 5 (12) | 12 (18) | 29 (41) | 21 (23)
Application site papules (General disorders) | 5 (5) | 4 (5) | 4 (4) | 1 (1) | 14 (14) | 13 (15)
Application site urticaria (General disorders) | 3 (3) | 9 (16) | 2 (3) | 1 (5) | 16 (34) | 5 (6)
Application site eczema (General disorders) | 7 (7) | 6 (7) | 5 (10) | 5 (5) | 14 (15) | 0 (0)
Application site erosion (General disorders) | 3 (3) | 2 (3) | 4 (4) | 1 (1) | 6 (8) | 11 (12)
Application site rash (General disorders) | 4 (5) | 3 (3) | 0 (0) | 1 (5) | 4 (5) | 2 (2)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 0 (0)
Application site vesicles (General disorders) | 0 (0) | 1 (3) | 3 (3) | 0 (0) | 2 (8) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 (32) | 10 (14) | 14 (46) | 20 (52) | 49 (114) | 37 (101)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (24) | 10 (22) | 7 (8) | 13 (22) | 19 (28) | 11 (21)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 6 (13) | 4 (4) | 2 (2) | 15 (25) | 19 (32)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (22) | 8 (10) | 5 (10) | 1 (1) | 11 (17) | 8 (22)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (14) | 2 (2) | 3 (8) | 7 (10) | 17 (34) | 3 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 10 (16) | 6 (7) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 3 (8) | 2 (2) | 3 (4) | 9 (14) | 5 (7)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 5 (6) | 1 (1) | 9 (9) | 5 (6)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (9) | 0 (0) | 2 (9) | 5 (6) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 18 (26) | 10 (11) | 15 (19) | 11 (18) | 45 (67) | 26 (31)
Hypersensitivity (Immune system disorders) | 10 (15) | 3 (3) | 10 (10) | 9 (16) | 33 (43) | 25 (40)
Food Allergy (Immune system disorders) | 7 (9) | 6 (10) | 4 (5) | 6 (8) | 22 (36) | 21 (30)
Seasonal allergy (Immune system disorders) | 6 (14) | 4 (5) | 3 (4) | 4 (4) | 17 (24) | 5 (11)
Allergy to animal (Immune system disorders) | 2 (3) | 4 (10) | 0 (0) | 0 (0) | 6 (11) | 9 (14)
Urticaria (Skin and subcutaneous tissue disorders) | 13 (24) | 14 (18) | 11 (25) | 7 (29) | 21 (30) | 17 (27)
Eczema (Skin and subcutaneous tissue disorders) | 11 (23) | 5 (7) | 9 (21) | 7 (16) | 24 (35) | 10 (12)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4) | 5 (5) | 4 (5) | 12 (20) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7) | 3 (7) | 2 (3) | 1 (1) | 7 (11) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (9) | 5 (5) | 5 (10) | 4 (6) | 18 (21) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 7 (9) | 0 (0) | 5 (6) | 4 (7) | 8 (9)
Oral pruritus (Gastrointestinal disorders) | 3 (4) | 1 (1) | 4 (5) | 4 (7) | 8 (9) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (4) | 4 (4) | 8 (9) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (4) | 2 (3) | 4 (6) | 5 (8)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 6 (7) | 3 (5)
Toothache (Gastrointestinal disorders) | 4 (7) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 5 (14) | 5 (8) | 5 (23) | 5 (6) | 12 (25) | 10 (27)
Eye swelling (Eye disorders) | 3 (10) | 2 (2) | 1 (1) | 0 (0) | 5 (7) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 5 (26) | 0 (0) | 1 (1) | 0 (0) | 5 (19) | 0 (0)
Application site oedema (General disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 10 (13) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT02223182/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT02223182/SAP_001.pdf